CLINICAL TRIAL: NCT06391788
Title: Efficacy and Safety of Thoracoscopic Morrow Surgery in the Treatment of Hypertrophic Obstructive Cardiomyopathy: a Single-center, Prospective, Open-label, Randomized, Controlled Trial
Brief Title: Efficacy and Safety of Thoracoscopic Morrow Surgery in the Treatment of Hypertrophic Obstructive Cardiomyopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-ZX013
Record Dates: First submitted 2024-04-15; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Cardiomyopathy, Hypertrophic Obstructive; Minimally Invasive Surgery
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracoscopic trans-mitral myectomy (Experimental): patients who undergo thoracoscopic Morrow procedure
  Interventions: Procedure: thoracoscopic Morrow surgery
- Modified extended Morrow myectomy (Active Comparator): patients who undergo modified extended Morrow myectomy
  Interventions: Procedure: modified Morrow surgery

INTERVENTIONS:
Procedure: thoracoscopic Morrow surgery — minimally invasive trans-mitral Morrow septal myectomy
  Arms: Thoracoscopic trans-mitral myectomy
Procedure: modified Morrow surgery — median open modified enlarged Morrow septal myectomy
  Arms: Modified extended Morrow myectomy

SUMMARY:
This single-center, prospective, open-label, randomized, controlled clinical trial is designed to assess the efficacy and safety of the Thoracoscopic Morrow procedure in the treatment of hypertrophic obstructive cardiomyopathy. The primary objectives include investigating:

Question 1: The efficacy and safety of two surgical modalities in patients presenting with left ventricular outflow tract obstruction and mid-left ventricular hypertrophy.

Question 2: The impact of the two surgical procedures on hemodynamics in patients with left ventricular outflow tract obstruction, mid-left ventricular obstruction, and in individuals with or without organic valvular lesions.

Question 3: The effects of the two surgical procedures on exercise capacity, quality of life, and long-term prognosis among patients with left ventricular outflow tract obstruction and central left ventricular obstruction, both with and without valvular lesions.

Participants will be stratified into two groups. The experimental group will undergo thoracoscopic Morrow surgery, while the control group will undergo median open modified enlarged Morrow surgery.

DETAILED DESCRIPTION:
This study is a single-center, prospective, open-label, randomized, controlled trial designed to investigate the therapeutic value of thoracoscopic Morrow procedure in patients with hypertrophic obstructive cardiomyopathy (HOCM). The study focuses on HOCM patients, with the modified extended Morrow procedure via median sternotomy considered as the 'gold standard treatment' in the control group. The objective is to explore the efficacy of the thoracoscopic Morrow procedure in improving exercise tolerance in HOCM patients, assess the short-term and long-term effectiveness, safety, as well as changes in cardiac function, cardiac structure, and myocardial fibrosis levels associated with thoracoscopic Morrow procedure in treating obstructive HOCM.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with hypertrophic cardiomyopathy (HCM);
* age ≥18 years old;
* presence of left ventricular outflow tract/mid-ventricular obstruction, with a resting left ventricular outflow tract pressure gradient/left ventricular cavity pressure gradient ≥50 mmHg; significant symptoms persist despite optimal medical therapy, and surgical evaluation indicates the need for intervention;
* left ventricular ejection fraction (LVEF) ≥55%;
* signed informed consent, willing and able to return to the hospital for follow-up.

Exclusion Criteria:

* previously underwent septal reduction therapy (including surgical or interventional procedures);
* received or planning to receive an implantable cardioverter-defibrillator (ICD) in the past 3 months;
* individuals with concomitant conditions requiring simultaneous surgical intervention;
* New York Heart Association (NYHA) functional class IV;
* unwilling to undergo surgical treatment;
* pregnant or lactating or planning pregnancy;
* previously participated in other clinical trials before enrollment;
* individuals with concurrent diseases with an expected lifespan of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular outflow tract gradient variability | 6 months,9 months and 12 months
  Change in Left ventricular outflow tract gradient pre- and post- intervention

SECONDARY OUTCOMES:
6-minute walk distance | 6 months,9 months and 12 months
  A measure used to assess the functional exercise capacity of individuals. It is determined by the distance a person can walk in 6 minutes on a flat, hard surface.
New York Heart Association Functional Classification of Heart Failure | 6 months,9 months and 12 months
  A system used to categorize the severity of heart failure based on the functional limitations of individuals.
Marker of myocardial injury | 6 months,9 months and 12 months
  To assay the concentration of proteins(cardiac troponin T, cardiac troponin I)associated with myocardial injury.
Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score | 6 months,9 months and 12 months
  A disease-specific health status measure designed to assess the impact of heart failure on patients' quality of life.
Echocardiographic indicator | 6 months,9 months and 12 months
  Left ventricular ejection fraction assessed by echocardiography.
Cardiac magnetic resonance indicator | 6 months,9 months and 12 months
  The left ventricular mass index was assessed using cardiac magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, Principal Investigator — Fuwai Hospital, National Centre for Cardiovascular Disease; Lei Song, Principal Investigator — Fuwai Hospital, National Centre for Cardiovascular Disease
Locations (1):
- Fuwai Hospital, National Centre for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No